CLINICAL TRIAL: NCT02804152
Title: A Novel Approach to Reduce Pain, Prescription Opioid Use & Misuse in Pregnancy
Brief Title: Program for Pain & Prescription Opioid Use in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1K23DA039318-01 (NIH)
Record Dates: First submitted 2016-05-10; First posted 2016-06-17 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Pain; Opioid Abuse; Pregnancy
Keywords: pregnancy; pain; prescription opioid
MeSH Terms: conditions — Pain; Opioid-Related Disorders | interventions — Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT for Chronic Pain (Other): single arm open-label design
  Interventions: Behavioral: CBT for Chronic Pain in Pregnancy

INTERVENTIONS:
Behavioral: CBT for Chronic Pain in Pregnancy — The content will be included in 8 weekly sessions, i.e., sessions 1-3 ("Education on chronic pain", "Theories of pain and diaphragmatic breathing" and "Progressive muscle relaxation and visual imagery"), sessions 4 and 5 ("Automatic thoughts and pain" and "Cognitive restructuring"), sessions 7, 8 and 10 ("Pleasant activity scheduling", "Time-based pacing" and "Sleep hygiene"), sessions 6 and 9 ("Stress management" and "Anger management"). Following this content, 1-2 sessions will be dedicated to review and reinforcement of key concepts or addressing any "stuck points" as well as cover content in session 11 ("Relapse Prevention"). The last session of therapy would include a review of achievements and commitment to continued application of CBT for chronic pain in participants daily lives.

SUMMARY:
Pregnant women using prescription opioid medication (pain medications) are invited to take part in a program for the reduction of pain and prescription opioid misuse.

DETAILED DESCRIPTION:
Subjects: Participants will be 200 adult, pregnant women receiving prenatal care and using POs for chronic pain. Women must be willing to consider a PO dose reduction, and cannot meet criteria for a Substance Use Disorder. Specific inclusion and exclusion criteria can be found in the Protections of Human Subjects section below.

Procedures: Pregnant women using POs will be identified by the obstetric care team, or self-referred via study advertisements, and referred to study personnel. The obstetric care team will serve as a referral source and will not be taking part in any research related activities. Women will be scheduled to meet with study personnel either in-person, via telemedicine or by phone and will undergo a brief eligibility screening. If women are eligible they will be given a full description of the study procedures and asked to read and sign an IRB-approved consent form in-person or consent online before any study procedures or assessments are conducted using doxyme software. Ineligible women, or those not wanting to take part will be referred for clinical treatment in-person or via telemedicine.

Baseline Visit: Eligible participants will complete online assessments (see primary outcome assessments below) via a Redcap survey. They will have their cell phones registered into the daily diary system described below and will be given instruction on how to respond to daily queries regarding pain, functioning, craving, mood etc. Participants without a cell phone will be provided a cell phone for use during the study. Eligible participants will complete daily ratings for no more than 21 days.

Treatment Phase: Immediately following the 21 day data collection phase, subjects will take part in 8, 75-minute sessions of the modified, individual CBT for Chronic Pain program. This treatment will be delivered once weekly over 8 weeks by the study therapist. Participants will continue their daily diary ratings and these will be reviewed by the study therapist and participant each week during the therapy session. Subjects will not receive any other CBT services during the study. All services received (e.g., pain management, self-help groups, case management) will be carefully monitored and tracked at weekly visits.

Each week, following the CBT for Chronic Pain session, the participant will meet with the study physician or APRN, for 15 minutes. PO use will be reviewed, symptoms of maternal or fetal withdrawal will be assessed (see Safety Measures and Appendix for medication management session) and based on the participant's preference, the provider will continue the same prescribed regime of the PO medication(s) or decrease the overall dose by 20%- a safe and recommended reduction of opioid medication during pregnancy14. Participant rational for their individual decision will be recorded and the appropriate amount of PO medication will be prescribed by the in-person provider or if via telemedicine, in collaboration with in-person obstetric provider. Use of POs from other providers will be carefully monitored and tracked at each weekly visit using the Prescription Drug Monitoring Program (PDMP) database and review of the EMR (see Safety Measures). Following each weekly treatment session, the participants will complete online assessments (see primary outcome assessments below) via a Redcap survey.

Follow-up: Women will be asked to continue their daily ratings for one month after completing the 8 week treatment. They will also be asked to complete an online assessment (see primary outcome assessments below) via a Redcap survey at one month post-treatment. At 6 weeks postpartum, women will be asked to complete their final online assessment (see primary outcome assessments below) via a Redcap survey.

ELIGIBILITY:
Inclusion Criteria:

* Adult females, any race or ethnicity, age 18-45 years.
* Pregnant and receiving prenatal care
* Willing to consider a decrease in their dose of their prescription opioid medication.
* Does not meet DSM-V criteria for a Substance Use Disorder.
* Able to comprehend English.
* Able to provide informed consent.

Exclusion Criteria:

* Unable to provide informed consent.
* Not currently pregnant, or receiving prenatal care
* Not currently taking a prescription opioid medication during pregnancy.
* Unwilling to consider a reduction in their prescription opioid medication dose.
* Meets DSM-V criteria for a Substance Use Disorder.
* Participation is not recommended by the participant's primary obstetrician

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) | change from baseline in BPI at 8 weeks, 1 month post treatment, and 6 weeks postpartum
  Pain Severity and Functioning
Current Opioid Misuse Measure (COMM) | change from baseline in COMM at 8 weeks, 1 month post treatment, and 6 weeks postpartum
  opioid misuse behaviors
Current Opioid Dose | change from baseline in current opioid dose at 8 weeks, 1 month post treatment, and 6 weeks postpartum
  Use of opioid medications in pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- The Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shapiro M, Sujan AC, Guille C. A Clinical Trial of a Program for Pain Management and Opioid Reduction During Pregnancy. Reprod Sci. 2022 Feb;29(2):606-613. doi: 10.1007/s43032-021-00701-4. Epub 2021 Aug 17. PMID 34403125